CLINICAL TRIAL: NCT03784378
Title: RXDX-105 for the Treatment of Patients With Non-Small Cell Lung Cancer (NSCLC) Harboring a RET Gene Fusion and a Patient With Ovarian Cancer Harboring a BRAF Gene Mutation
Brief Title: Continued Access to RXDX-105
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-487
Record Dates: First submitted 2018-12-17; First posted 2018-12-21 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2020-09

CONDITIONS: Non Small Cell Lung Cancer; Ovarian Cancer; RET Gene Mutation; BRAF Gene Mutation
Keywords: RXDX-105; Memorial Sloan Kettering Cancer Center; 18-487
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms | interventions — agerafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants previously enrolled on Study of RXDX-105 (Experimental): Participants were previously enrolled on Study of RXDX-105
  Interventions: Drug: RXDX-105

INTERVENTIONS:
Drug: RXDX-105 — RXDX-105 capsules will be administered orally on a continuous daily dosing regimen. Patients will be continue to be treated at the dose level they were previously treated on during participation on Study of RXDX-105.

SUMMARY:
This study is being done to see if people with Non-Small Cell Lung Cancer (NSCLC) or ovarian cancer benefit from continued treatment with the study drug, RXDX-105.

ELIGIBILITY:
Inclusion Criteria:

* This individual patient protocol includes treatment for 3 patients previously enrolled on IRB #15-270 (phase1/1b clinical trial RXDX-105-01):

Exclusion Criteria:

* Any patients other than those described above are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluation during treatment/intervention | Through study completion, up to five years.
  Safety assessments will be performed as standard of care and as clinically indicated. This will include monitoring of adverse events, including serious adverse events including CTCAE grading.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Drilon, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center 1275 York Avenue, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org